CLINICAL TRIAL: NCT04652427
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Clinical Trial Program on the Effectiveness and Safety of Dexmedetomidine Hydrochloride Injection for Sedation in Patients Without Tracheal Intubation
Brief Title: Application of Dexmedetomidine Hydrochloride Injection in Anesthesia for Patients Without Tracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Director of department of anesthesiology and pain management, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020PHC003
Record Dates: First submitted 2020-08-20; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Sedation Complication
Keywords: effectiveness; security; Dexmedetomidine Hydrochloride; Non-tracheal intubation anesthetic
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Use Dexmedetomidine Hydrochloride to maintain a sedative (Experimental): Slow static injection at a load-loaded dose of 1.0/g/kg (half of the load dose in ophthalmology surgery), infusion time of 10 to 15 min, followed by the maintenance phase, maintenance dose set at an initial 0.6/g/kg/h, maintenance during administration The researchers, using the results of the OAA/S assessment, made a comprehensive judgment to adjust the infusion rate in the range of 0.2 to 1.0/g/kg/h to obtain the desired sedative effect, and anaesthetic can be performed when the study drug was given a duration of 15 minutes and the required sedative level was reached. Maintain the administration until the end of the operation.
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.1 MG/ML
- Sedative were maintained with a 0.9% sodium chloride injection (Placebo Comparator): Slow static injection at a load-loaded dose of 1.0/g/kg (half of the load dose in ophthalmology surgery), infusion time of 10 to 15 min, followed by the maintenance phase, maintenance dose set at an initial 0.6/g/kg/h, maintenance during administration The researchers, using the results of the OAA/S assessment, made a comprehensive judgment to adjust the infusion rate in the range of 0.2 to 1.0/g/kg/h to obtain the desired sedative effect, and anaesthetic can be performed when the study drug was given a duration of 15 minutes and the required sedative level was reached. Maintain the administration until the end of the operation.
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride 0.1 MG/ML — At least 15 min prior to anesthesia is sedated by the study drug given according to the administration protocol, an alert/sedative score (OAA/S) is performed at the end of the drug load dose administration, and then the maintenance-giving phase is then performed at the end of the operation with an OAA/S score every 5 min. Anestheticing can be performed after the required level of sedation has been reached. OAA/S 4 should always be maintained during drug administration.
  Other Names: sedation
  Arms: Use Dexmedetomidine Hydrochloride to maintain a sedative
Drug: 0.9% Sodium Chloride Injection — At least 15 min prior to anesthesia is sedated by the study drug given according to the administration protocol, an alert/sedative score (OAA/S) is performed at the end of the drug load dose administration, and then the maintenance-giving phase is then performed at the end of the operation with an OAA/S score every 5 min. Anestheticing can be performed after the required level of sedation has been reached. OAA/S 4 should always be maintained during drug administration.
  Other Names: saline solution
  Arms: Sedative were maintained with a 0.9% sodium chloride injection

SUMMARY:
With 0.9% sodium chloride injection as a placebo control, to evaluate the effectiveness and safety of dexmedetomidine hydrochloride injection for sedation in patients with non-tracheal intubation

DETAILED DESCRIPTION:
Clinically common non-systemic anesthesia mainly includes surface anesthesia, local immersion anesthesia, nerve block, regional blocking, intravertebral anesthesia. Patients under non-general anesthesia surgery, is still in a more sober state, easily due to external factors and increase the psychological and mental burden, even if the ideal anaesthetic effect can be achieved, but for autonomic nerve activities can not be completely and effectively eliminated. Hydrochloric acid right-metomidine is an alpha2-adrenaline receptor agonisant developed by Orion Pharma (Finland) and Abott (Usa) in collaboration. Unlike other sedative hypnotic sedatives, hydrochloric acid right metamine produces a sedative hypnotic effect by acting on the blue spot nuclear alpha2 receptor and the inflammatory endogenous sleep-stimulating pathway, allowing the patient to maintain a natural sleep state of non-fast eye III, which is characterized by the patient being stimulated or speech-altered, and does not produce respiratory inhibition during sedative hypnosis. In addition to the sedative effect, the right metomisurein also has anti-anxiety, reduce stress response, stable hemodynamics, analgesic, inhibitsalival secretion, anti-cold and diuretic function, and other sedative analgesic drugs when used with good synergy, can significantly reduce the use of other sedative analgesic drugs.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18~65 years old (including 18 and 65 years old), no gender limit;
* 2) 18 kg/m2 ≤BMI≤30 kg/m2;
* 3) For patients undergoing elective surgery under non-general anesthesia, the expected duration of surgery is ≥30min;
* 4) ASA classification is Ⅰ～Ⅲ;
* 5) After the patient has a full understanding of the purpose and significance of this trial, he/she voluntarily participates in this clinical trial, agrees to contraception during the study period and within 3 days after the study medication, and signs an informed consent Intent.

Exclusion Criteria:

* 1) Patients who have received anesthesia or surgery within 7 days before randomization;
* 2) Patients with a history of acute myocardial infarction or unstable angina within 6 months before the screening period;
* 3) Bradycardia (heart rate <50 beats/min), Ⅱ or Ⅲ degree atrioventricular block (not including Patients with pacemakers) and other severe arrhythmia and heart failure;
* 4) Hypertension patients who are not satisfactorily controlled (systolic blood pressure ≥160 mmHg, and/or diastolic blood pressure ≥100 mmHg), or patients with hypotension (systolic blood pressure <90 mmHg);
* 5) People with mental system diseases (such as schizophrenia, depression, etc.) or cognitive impairment; Those with a history of epilepsy;
* 6) Those who suffer from bronchial asthma or other severe respiratory diseases;
* 7) Abnormal blood coagulation function (PT prolongation exceeds the upper limit of normal for 3 seconds and/or APTT prolongation exceeds. The upper limit of the normal value is 10 seconds);
* 8) Abnormal liver and kidney function (ALT and/or AST>2 times the upper limit of normal, total bilirubin>1.5 Times the upper limit of normal, blood creatinine>1.5 times the upper limit of normal);
* 9) Those who have used α2 adrenergic receptor agonists or antagonists within 14 days before randomization;
* 10) Those who have used sedatives such as benzodiazepines and barbiturates within 7 days before randomization;
* 11) People with a history of drug abuse, drug abuse and alcohol abuse, among which alcohol abuse is defined as the average daily drinking Liquor exceeds 2 units of alcohol (1 unit = 360 ml of beer or 45 ml of alcohol is 40% white wine or 150 ml wine);
* 12) Those who are allergic to dexmedetomidine, midazolam, fentanyl and other pharmaceutical ingredients or components;
* 13) Women who are pregnant or breastfeeding;
* 14) Those who have participated in other clinical trials within 3 months before randomization;
* 15) The researcher believes that there are any other circumstances that are not suitable for selection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the OAA/S score of the subject during the study medication. | 15min after giving the drug, every five minutes during anesthesia
  At least 15 minutes before anesthesia, the study drug was given sedation according to the dosing schedule. At the end of the loading dose of the study drug, an alertness/sedation score (OAA/S) was performed, and then it entered the maintenance dosing phase, which was performed every 5 minutes until the end of the operation OAA/S score. OAA/S≤4 means that the required level of sedation has been reached, and anesthesia can be performed after starting the study drug for ≥15 minutes and reaching the required level of sedation. During the administration of the study drug, OAA/S ≤4 should always be maintained.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Feng, MD,PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Candiotti KA, Bergese SD, Bokesch PM, Feldman MA, Wisemandle W, Bekker AY; MAC Study Group. Monitored anesthesia care with dexmedetomidine: a prospective, randomized, double-blind, multicenter trial. Anesth Analg. 2010 Jan 1;110(1):47-56. doi: 10.1213/ane.0b013e3181ae0856. Epub 2009 Aug 27. PMID 19713256